CLINICAL TRIAL: NCT04790188
Title: Effect of a Nootropic on the Cognitive Performance in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Jonatan Ruiz Ruiz, Associate professor, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: NOCOPE project
Record Dates: First submitted 2021-03-03; First posted 2021-03-10 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Cognitive Change
MeSH Terms: interventions — Nootropic Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental intervention first. (Experimental): Participants randomized to receive the nootropic first.
  Interventions: Dietary Supplement: Nootropic; Dietary Supplement: Placebo
- Experimental intervention second. (Placebo Comparator): Participants randomized to receive the placebo first
  Interventions: Dietary Supplement: Nootropic; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nootropic — 10g of Evo-Gamers® lemon flavor (HSN®). The nutritional composition per service is: L-Tyrosine (1000mg), Acetyl L-Carnitine HCL (500mg), Citicoline sodium (200mg), L-alpha-Glycerylphosphorylcholine (Alpha-GPC; 100mg), Vitamin C (150mg), Vitamin E (12.1mg), Vitamin B6 (3mg), Vitamin B2 (3mg), Vitamin A (810μg), Vitamin D (10μg), Vitamin B12 (5μg), Taurine (500mg), Caffeine (300mg), L-Theanine (150mg), Mango Leaves (2000mg), Huperzia Leaves (200mg). The dose to be administered is that recommended on the labeling and nutritional information of the nootropic which has been produced under GMP procedures and approved by the EFSA.
Dietary Supplement: Placebo — 10g of maltodextrin lemon flavor (HSN®).

SUMMARY:
The main aim of this study is to determine the effect of a nootropic on cognitive performance (i.e., reaction time, inhibitory control, cognitive flexibility, working memory, neuro-psychological outcomes).

DETAILED DESCRIPTION:
Cognitive decline is a worrisome consequence of normal or pathologic ageing, having a high personal, eco- nomic and societal burden; also, it could herald the onset of dementia which is associated with significant morbidity and mortality.

However, with a general increase in life expectancy and a corresponding increase in the prevalence of age-related cognitive impairment, there have been concerted efforts towards the development and adoption of preventive strategies that would minimize the risk of developing dementia, or reduce the rate of cognitive decline with ageing. In the last few decades, certain compounds have been found useful in the management of cognitive decline.

The term 'nootropic' has been used to define such substances with the capacity to enhance cognition. While research has led to the synthesis of several drugs with nootropic effects, attention is now being shifted to the discovery, characterization and utilization of nootropics from natural sources for the prevention and management of age-related cognitive decline.

25 young adults will be randomized into two conditions (nootropic and placebo conditions) with 48 hours of separation between conditions. 48h previous to the randomization the participants will perform a familiarization to avoid the learning effects.

Each evaluation day will conform to the following tests:

* Simple and multiple reaction time
* Inhibitory control
* Cognitive flexibility
* Working memory
* Creative intelligence
* Verbal fluidity
* Motivation
* Mood
* Positive and negative emotions
* Adverse effects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Ages 18-30 years
* BMI: 18-30.0 kg/m2
* Stable weight over the last 3 months (body weight changes<3kg)
* Participant must be capable and willing to provide consent, understand exclusion criteria, instructions and protocols.
* To talk and to read Spanish fluently.

Exclusion Criteria:

* History of neurological disease or mental disease.
* History of cardiovascular disease
* Diabetes or hypertension
* Pregnant, planning to become pregnant, or breastfeeding
* Have been treated previously or during the study period with neurological drugs.
* Have been treated previously or during the study period with prescription drugs: antihypertensive, lipid lowering, acid uric lowering, glucose lowering, beta blockers or any drug that under the investigator's judged could influence the results.
* Allergy/intolerance to any ingredient of the nootropic.
* High caffeine consumes (>300mg/day, or >3 coffees/day).
* Any non-controlled medical condition which could influence results or could be worsened by the participation in the study.
* Are deemed unsuitable by the investigator for any other reason, that prevent data collection.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Simple and multiple reaction time | 1.5 hours
  Vienna Test System®

SECONDARY OUTCOMES:
Inhibitory control | 1.5 hours
  Stroop test, E-Prime® software
Working Memory | 1.5 hours
  Tests Flankers and Task switching, EPrime ® software
Working memory | 1.5 hours
  N-Back y Spatial working memory , EPrime ® software
Creative Intelligence | 1.5 hours
  CREA test
Verbal fluidity | 1.5 hours
  Phonological and semantic verbal fluidity
Motivation | 1.5 hours
  Situational Motivation Scale (EMSI)
Mood | 1.5 hours
  EVEA scale
Positive and negative emotions | 1.5 hours
  PANAS scale
Adverse effects | 1.5 hours
  Visual analogue scales of adverse effects (gastrointestinal, nervous or psychologic)

CONTACTS AND LOCATIONS:
Locations (1):
- Jonatan Ruiz Ruiz, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Medrano M, Molina-Hidalgo C, Alcantara JMA, Ruiz JR, Jurado-Fasoli L. Acute Effect of a Dietary Multi-Ingredient Nootropic as a Cognitive Enhancer in Young Healthy Adults: A Randomized, Triple-Blinded, Placebo-Controlled, Crossover Trial. Front Nutr. 2022 May 12;9:858910. doi: 10.3389/fnut.2022.858910. eCollection 2022. PMID 35634417